CLINICAL TRIAL: NCT04071873
Title: A Novel Approach to Community-based HIV Testing With Traditional Healers in Mwanza, Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-04020274
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-10

CONDITIONS: HIV; Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Point-of-care HIV testing (intervention) (Experimental): Participants will be offered voluntary point-of-care HIV testing during a traditional healer visit.
  Interventions: Diagnostic Test: Point-of-care HIV testing
- Education on community HIV resources (control) (Active Comparator): Participants will be offered education regarding HIV testing and community resources during a traditional healer visit.
  Interventions: Behavioral: HIV testing education

INTERVENTIONS:
Diagnostic Test: Point-of-care HIV testing — Participants will undergo an HIV 1/2 antibody point of care test (Oraquick) and receive pre- and post-test counselling.Participants with positive tests will be referred to the HIV clinic for Western Blot confirmation, and linkage to care.
  Arms: Point-of-care HIV testing (intervention)
Behavioral: HIV testing education — Participants will be provided with education on community based HIV resources.
  Arms: Education on community HIV resources (control)

SUMMARY:
HIV antiretroviral therapy (ART) has the potential to dramatically decrease HIV transmission worldwide. In Tanzania, HIV prevalence is ~5%, with 1.6 million people living with HIV/AIDS; it is the leading cause of hospitalization and death among Tanzanian adults. However, less than 50% of HIV-infected Tanzanian adults know their status.Successful implementation of community-based services requires an understanding of the social and cultural context that influence community engagement with HIV services. Specifically, many HIV endemic regions are also medically pluralistic communities, where multiple explanatory frameworks for health and disease co-exist. In these areas, HIV testing and ART clinical care do not occur in isolation; traditional healers are commonly utilized instead of or concurrently with biomedical services. Therefore, the success of decentralized, community-based HIV services must be founded upon a thorough understanding of medical pluralism, and engagement with traditional healers as stakeholders in community health.

This study will investigate the feasibility of involving traditional healers in HIV testing, and pilot an intervention to expand HIV testing within communities that use traditional medicine in Mwanza, Tanzania.

DETAILED DESCRIPTION:
This study has two specific aims.

Specific Aim 1:

Tailor a point of care HIV testing intervention for delivery in northwestern Tanzania, using data from 1) qualitative interviews and 2) community engagement strategies. Interviews with traditional healers, traditional and biomedical clients, and HIV clinic staff will illustrate local variables impacting HIV testing engagement. A community advisory board with stakeholder members will guide program implementation, tailoring protocols to maximize uptake.

Specific Aim 2:

Conduct a cluster-randomized pilot of the HIV testing intervention. This pilot will offer HIV testing at five traditional healer practice sites, compared with a control group of five healers providing education on community HIV resources..

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Not known to be HIV-infected
* Client of a traditional healer practice
* Willing to be contacted for monthly follow-up for three months
* Willing to complete an exit survey at the end of three months
* Able to provide informed consent

Inclusion specific to point-of-care HIV testing intervention:

* Willing to have point of care HIV test
* Willing to receive results of HIV test

Exclusion Criteria:

* less than 18 years of age
* Known to be HIV-infected
* Unable to provide informed consent
* Unwilling to participate in follow-up

Exclusion specific to point-of-care HIV testing intervention:

* Unwilling to have point-of-care HIV test
* Unwilling to receive the results of HIV test

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of HIV testing | Within 3 months following visit
  Rate of HIV testing among clients of traditional healers who were offered point-of-care HIV testing, as compared to clients who were offered education regarding community HIV resources.

SECONDARY OUTCOMES:
Rate of new HIV diagnosis | 3 months
  Rate of new HIV diagnosis among clients of traditional healers who were offered point-of-care HIV testing, as compared to clients who were offered education regarding community HIV resources.

OTHER OUTCOMES:
Linkage to HIV care at 3 months post enrollment | 3 months
  Rate of successful care linkage for participants with a new HIV diagnosis who received point-of-care HIV testing as compared to participants who received education regarding community HIV resources.Linkage to care will be defined as accessing outpatient care or treatment such as antiretroviral therapy (ART).

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Sundararajan, PhD, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- National Institute for Medical Research, Mwanza, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be made available.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication.
Access Criteria: Requests should be directed to ras9199@med.cornell.edu .